CLINICAL TRIAL: NCT06879301
Title: Effectiveness of Intravitreal Injection of Aflibercept 8 mg in Resistant Diabetic Macular Edema and Retinal Vein Occlusion Patients
Brief Title: Effectiveness of Intravitreal Injection of Aflibercept 8 mg in Resistant Diabetic Macular Edema, Retinal Vein Occlusion and Myopic Choroidal Neovascularisation Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amin El Sayed Nawar, Associate professor of ophthalmology, Tanta University,Egypt, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEN; Tanta university (Other: Tanta University)
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Macular Edema (DME); Retinal Vein Occlusion (RVO); Myopic Choroidal Neovascularisation
Keywords: Aflibercept 8 mg; diabetic macular edema
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 60 eyes of resistant diabetic macular edema (Experimental): This prospective interventional case study will be conducted on 60 eyes of 60 patients with resistant centrally involved diabetic macular edema following at least 3 doses of anti_VEGF therapy including cases receive previous injection of ranibzumab and aflibercept 2 mg.
  All procedures were carried out under the tenets of the Helsinki Declaration. Written consent was provided by all participants after discussing the procedure, alternative treatment plans, follow-up schedules, and possible benefits and risks.
  Participants: This study included resistant centrally involved diabetic macular edema (DME) cases
  Interventions: Drug: Intravitreal injection of aflibercept 8 mg

INTERVENTIONS:
Drug: Intravitreal injection of aflibercept 8 mg — Preoperative preparation: Patients were prepared by applying topical fluoroquinolone eye drops (moxifloxacin hydrochloride 0.5% Vigamox, Alcon, USA) 4 times daily for three days before injection.
  Procedure: The intravitreal injection was carried out in the operating room under complete aseptic techniques with an operating microscope. After the topical application of anaesthetic drops (benoxinate hydrochloride 0.4%, Benox, Epico, Egypt) to the ocular surface followed by the topical application of 10% povidone-iodine (Betadine) to the periocular area, lids and eye lashes, 5% povidone iodine was administered inside the conjunctival sac for three minutes before the intravitreal injection. 0.07 ml of aflibercept (8 mg) was injected into the vitreous cavity in the inferotemporal quadrant of the globe using a 30-gauge needle 4 mm from the limbus.
  Postoperative care: After injection, topical antibiotic drops (moxifloxacin hydrochloride 0.5% Vigamox, Alcon, USA) were applied, and the eye was

SUMMARY:
Generally, DM is caused by insufficient insulin secretion in the body; however, the other biological mechanisms remain unclear. Long-term illness in patients with DM damages various organs in the body, such as the eyes, kidneys, and heart, seriously affecting organ function. Nowadays, the quality of life of people has improved significantly, eating habits have changed, sugar intake is increasing, and the number of patients with DM is increasing. Statistics show that in 2017, the number of patients with DM worldwide reached 425 million (aged 20-79 years), which will exceed 600 million in 30 years; moreover, patients in low- and middle-income countries, such as China and India, account for 80 percent of the total DM population (1). According to the WHO, patients with DM worldwide increased to 366 million in 2011, which is expected to increase to 500 million in 2025, with more than 150 million patients experiencing ocular complications, such as diabetic retinopathy (DR) (2, 3). DR is a form of ocular microangiopathy and the most serious DM-related complication; it seriously endangers the health of patients with DM (4). DR pathogenesis includes increased endothelial cells in the eye capillaries, increased intimal thickness, damaged pericytes, microangioma, and damaged blood-retina barrier due to increased permeability of the blood vessels, microvascular obstruction, and neovascularization (NV) (5, 6). Currently, the prevalence of DR is 34.6% worldwide; however, it is higher in some developed countries, reaching 40.3% (7). The proportion of patients with type 1 and 2 DM suffering from blindness due to DR is 3.6% and 1.6%, respectively (8). DR is associated with significantly reduced living standards, huge medical costs, and increased social burden (9, 10).

Many anti-vascular endothelial growth factor (VEGF) drugs exist; however, the use of therapeutic drugs is strictly controlled. The main drugs recommended for treating DM-related visual complications are ranibizumab and aflibercept.

DETAILED DESCRIPTION:
Study design: This prospective interventional case study will be conducted on 60 eyes of 60 patients with resistant centrally involved diabetic macular edema following at least 3 doses of anti_VEGF therapy including cases receive previous injection of ranibzumab and aflibercept 2 mg.

All procedures were carried out under the tenets of the Helsinki Declaration. Written consent was provided by all participants after discussing the procedure, alternative treatment plans, follow-up schedules, and possible benefits and risks.

Participants: This study included resistant centrally involved diabetic macular edema (DME) cases Patients with a history of intraocular surgery, coincident retinal pathology such as retinal vascular occlusion, CNV due to age-related macular degeneration, angioid streaks, trauma, and choroiditis were excluded from the study. In addition, patients who received other lines of treatment for DME, such as laser photocoagulation, intravitreal injecrion of steroids and patients known to be glaucomatous or have an IOP ≥20 mmHg were also excluded.

Furthermore, patients with other retinal pathologies, such as prior ocular inflammation, retinal degeneration, and dense media opacity, including nuclear sclerosis, and those who did not complete 1 year of follow-up were not enrolled in the present study.

A thorough ophthalmic evaluation, including a BCVA test using a Snellen chart that was converted to LogMAR for statistical analysis, IOP measurements using applanation tonometry, an anterior segment examination using a slit lamp, a posterior segment examination by slit lamp bimicroscopy using a +78 D lens, and indirect ophthalmoscopy, was performed for all patients. Spectral-domain OCT (Topcon 3D Optical Coherence Tomography) was performed for all patients at baseline and at the postoperative first-month visit and then monthly for 1 year.

Surgical procedure:

Preoperative preparation: Patients were prepared by applying topical fluoroquinolone eye drops (moxifloxacin hydrochloride 0.5% Vigamox, Alcon, USA) 4 times daily for three days before injection.

Procedure: The intravitreal injection was carried out in the operating room under complete aseptic techniques with an operating microscope. After the topical application of anaesthetic drops (benoxinate hydrochloride 0.4%, Benox, Epico, Egypt) to the ocular surface followed by the topical application of 10% povidone-iodine (Betadine) to the periocular area, lids and eye lashes, 5% povidone iodine was administered inside the conjunctival sac for three minutes before the intravitreal injection. 0.07 ml of aflibercept (8 mg) was injected into the vitreous cavity in the inferotemporal quadrant of the globe using a 30-gauge needle 4 mm from the limbus.

Postoperative care: After injection, topical antibiotic drops (moxifloxacin hydrochloride 0.5% Vigamox, Alcon, USA) were applied, and the eye was patched for several hours. Patients were instructed to administer antibiotic drops four times daily for 3 days. Patients were examined the following day and the third day after injection to exclude any complications, such as an elevated IOP, endophthalmitis, retinal breaks, retinal detachment and vitreous hemorrhage. All patients were followed up at 4-week intervals after the first injection. At each visit, a thorough ophthalmic examination and SD-OCT were performed. Pro re nata (PRN) regimen was followed in this study, in which an additional intravitreal injection will be given monthly if no improvement in or stabilization of best corrected visual acuity (improvement by more than one line in the Snellen chart) and/or persistent neurosensory detachment was detected on SD-OCT.

ELIGIBILITY:
Inclusion Criteria:

This study included resistant centrally involved diabetic macular edema (DME) cases

-

Exclusion Criteria:

1. Patients with a history of intraocular surgery
2. coincident retinal pathology such as retinal vascular occlusion, CNV due to age-related macular degeneration, angioid streaks, trauma, and choroiditis were excluded from the study.
3. patients who received other lines of treatment for DME, such as laser photocoagulation, intravitreal injection of steroids
4. patients known to be glaucomatous or have an IOP ≥20 mmHg were also excluded.

   -

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-19 (Estimated); Primary Completion 2025-11-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity | 1 MONTH
  improvemnt of BCVA after intravitrreal injection of eylea HD

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No